CLINICAL TRIAL: NCT01121978
Title: Early Vitrectomy for Macular Tractional Maculopathy. Multicenter Clinical Trial
Brief Title: Early Vitrectomy for Macular Tractional Maculopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul Retina Investigator Group (Network)
Responsible Party: Se Woong Kang, Samsung Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SRIG #2
Record Dates: First submitted 2010-04-30; First posted 2010-05-12 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2011-03

CONDITIONS: Myopia, Degenerative
Keywords: macular tractional maculopathy; pathologic myopia
MeSH Terms: conditions — Myopia, Degenerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conservative treatment group (No Intervention): Eyes which do not undergo early vitrectomy at the time of enrollment. Surgical intervention would be performed when full-thickness macular hole or vision deterioration occurs
- Early vitrectomy (Experimental): Triamcinolone acetonide assisted pars plana vitrectomy with Indocyanine green dye assisted internal limiting membrane peeling
  Interventions: Procedure: Early vitrectomy

INTERVENTIONS:
Procedure: Early vitrectomy — Triamcinolone acetonide assisted pars plana vitrectomy with Indocyanine green dye assisted internal limiting membrane peeling
  Other Names: pars plana vitrectomy for macular tractional maculopathy
  Arms: Early vitrectomy

SUMMARY:
This study is designed to identify the effect of current vitreous surgery for symptomatic macular tractional maculopathy.

Characteristics of this study is as below

1. Multicenter, prospective clinical trial. (early surgical intervention vs.surgical intervention when full-thickness macular hole formation or deterioration of visual acuity occurs)
2. Non-randomized study (decision was made by patients after full explanation)
3. After 1 year follow up, functional change(visual acuity)and anatomical change would be evaluated

DETAILED DESCRIPTION:
Degenerative myopia is relatively common disorder, especially in Korean, Japanese and Chinese.

Choroidal neovascularization is well-noted cause of VA deterioration, but nowadays, with improvement of diagnostic tools, such as OCT, VA deterioration from myopic tractional maculopathy is being concerned as well.

But till now, the necessity of early vitrectomy on MTM is controversial. By now some clinicians prefer conservative treatment, which means pars plana vitrectomy would be postponed till structural change such as macular hole formation is noticed. And the others prefer early vitrectomy, which means pars plana vitrectomy should be performed when the symptom begins.

In this study, investigators try to verify the validity of early vitrectomy comparing conservative treatment.

ELIGIBILITY:
Inclusion Criteria:

* male or female with impending macular hole(identified with OCT)
* Age: over 20 years
* Symptom duration < 6 Months
* Visual acuity on trial: more than 20/320 in ETDRS chart

Exclusion Criteria:

* Any vision disturbing disease other than impending macular hole
* Diabetic maculopathy or other retinal vascular disease
* Prior history of major trauma: If symptom begins after trauma
* Any evidence of atrophic change, scar or exudation on macula active intraocular inflammation
* History of intraocular surgery other than uncomplicated cataract extraction 3 months before
* Uncontrolled IOP > 25mmHg

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual acuity | 48 weeks

SECONDARY OUTCOMES:
Rate of occurrence of full-thickness macular hole | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Se Woong Kang, M.D., Principal Investigator — Seoul Retina Investigator Group
Locations (10):
- South Korea (10):
  - Asan Medical Center, University of Ulsan College of Medicine, Seoul, 82-2-3010-3673
  - Konyang University, Myung Gok Eye Research Institute, Daejeon, Daejeon
  - Seoul National University Bundang Hospital, Seongnam, Gyunggi-do
  - HanGil Eye Hospital, Incheon, In Cheon
  - Seoul National University Hospital, Seoul, Seoul
  - Kangdong Sacred Heart Hospital, Hallym University College of Medicine,, Seoul, Seoul
  - Samsung Medical Center, Seoul, Seoul
  - Catholic University of Korea, Seoul, Seoul
  - Gangnam Sacred Heart Hospital,Hallym University, Seoul, Seoul
  - Kong eye clinic, Seoul, Seoul